CLINICAL TRIAL: NCT00951873
Title: A Single-centre, Randomised, Placebo-controlled, Double-blind Single Dose, Dose Escalation Trial Investigating Safety, Pharmacokinetics and Local Tolerability of Ascending Subcutaneous Doses of Long Acting-rFVIIa in Healthy Male Subjects
Brief Title: A Single Dose Trial Investigating Safety and Local Tolerability of Ascending Doses of Long Acting Activated Recombinant Human Factor VII in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN7129-3754; 2009-011267-37 (EudraCT Number)
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Haemophilia B; Healthy
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: activated recombinant human factor VII, long acting
- B (Placebo Comparator)
  Interventions: Drug: placebo
- C (Experimental)
  Interventions: Drug: activated recombinant human factor VII, long acting

INTERVENTIONS:
Drug: activated recombinant human factor VII, long acting — Single injection of long acting activated recombinant human factor VII subcutaneously (under the skin). Each treatment dose of 0,1 mg/kg, 0,3 mg/kg and 0,5 mg/kg is assessed for safety before escalating to next dose.
  Arms: A
Drug: placebo — Single injection of long acting activated recombinant human factor VII placebo subcutaneously (under the skin). Each treatment dose of 0,1 mg/kg, 0,3 mg/kg and 0,5 mg/kg is assessed for safety before escalating to next dose.
  Arms: B
Drug: activated recombinant human factor VII, long acting — Single dose of 0,1 mg/kg long acting activated recombinant human factor VII injected intravenously (into a vein).
  Arms: C

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to investigate the safety, local tolerability and pharmacokinetic profile (the determination of the concentration of the administered medication in blood over time) of long acting activated recombinant human factor VII when injected subcutaneously (under the skin).

ELIGIBILITY:
Inclusion Criteria:

* Caucasian origin
* Body weight between 50 and 100 kg and a Body Mass Index (BMI) between 18.0 and 28.0 kg/m2 inclusive
* Smoke less than 10 cigarettes/day or equivalent and willingness to abstain from smoking during the entire duration of Trial Product Administration (9 days)

Exclusion Criteria:

* Known or suspected allergy to trial product or related products, such as activated recombinant human factor VII (NovoSeven®)
* Previous participation in this trial, defined as randomised to receive trial product
* Evidence of clinically relevant pathology or potential thromboembolic risk as judged by the Investigator
* Known history of atherosclerosis or thromboembolic events
* Overt bleeding, including from gastrointestinal tract
* Hepatitis B or C infection
* HIV infection
* Positive test for drugs of abuse

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2009-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | assessed throughout the trial period from visit 1 to visit 5

SECONDARY OUTCOMES:
Area under activity concentration-time curve from time zero to infinity | assessed up to 168 hours after trial product administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Harrow, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com